CLINICAL TRIAL: NCT01417793
Title: Effects of a Smoking Cessation Program for Prison Inmates-A Case Study of a Prison in Central Taiwan
Brief Title: Effects of a Smoking Cessation Program for Prison Inmates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Yulung Chen, China Medical University Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: DMR100-IRB-129
Record Dates: First submitted 2011-08-14; First posted 2011-08-16 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation rate
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Smoking Cessation Program (Experimental)
  Interventions: Behavioral: Smoking Cessation Program

INTERVENTIONS:
Behavioral: Smoking Cessation Program — Comparison of smoking cessation rate among different smoking cessation program

SUMMARY:
According to WHO database, an average of 540 million people worldwide dies from smoking related diseases every year. The use of tobacco products may reduce the average life expectancy of about 15 years. The data of 2009 from Department of Health Bureau of Health showed 38.57% male adults and 4.75% female adults smoked in Taiwan. Studies about smoking rate within prison inmates were between 64-91.8%, which was over 3 times than the general population. Smoking cessation can lower the risks of smoking related health problems. Two thirds of smokers in Taiwan once tried smoking cessation but the success rate was about 5% every year.

In view of high smoking rate within prison inmates in Taiwan, Agency of Correction, Ministry of Justice announced a smoking cessation program for inmates in April 2010. The purpose of this study was to investigate the effects of this program and the difference of cessation success rate between various interventional methods, using questionnaires for smokers and smoking cessation clinics database.

ELIGIBILITY:
Inclusion Criteria:

* Prison inmates with age equal or more than 20 years old and have smoked for equal or more than one year

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-08; Primary Completion 2012-05 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Smoking Cessation Rate | 6 months after each subject's enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Yulung Chen, M.D, Principal Investigator — China Medical University Hospital
Locations (1):
- Taichung Prison,Agency of Corrections, Ministry of Justice, Taichung, Taiwan, Taiwan